CLINICAL TRIAL: NCT02836990
Title: Prevena™ Incision Management System Versus Dermabond in the Prevention of Groin Wound Infections in Patients Undergoing Vascular Surgery
Brief Title: Prevena™ vs Dermabond in Groin Wound Infections in Vascular Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: KCI USA, Inc (Industry)
Responsible Party: Principal Investigator, Linda Harris, Professor, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Prevena
Record Dates: First submitted 2016-07-11; First posted 2016-07-19 (Estimated); Results first posted 2020-12-28 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Wound Infection
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prevena (Active Comparator): Prevena Incision Management System for vascular surgical groin wounds
  Interventions: Device: Prevena Incision Management System
- Dermabond (Active Comparator): Dermabond for vascular surgical groin wounds
  Interventions: Device: Dermabond

INTERVENTIONS:
Device: Prevena Incision Management System — A negative pressure system which holds incision edges together and removes exudate and debris from site to prevent surgical wound infections
  Other Names: Prevena
  Arms: Prevena
Device: Dermabond — A surgical skin adhesive used to prevent surgical wound infections
  Arms: Dermabond

SUMMARY:
This study evaluates the clinical efficacy and cost effectiveness of Prevena Incision Management System versus Dermabond in preventing groin wound infections in patients who undergo vascular surgery requiring a groin wound. Half of the patients will receive Dermabond and the other half will receive the Prevena Incision Management System for their groin wounds.

DETAILED DESCRIPTION:
Dermabond and the Prevena Incision Management System are both FDA approved wound care products. Prevena is a negative pressure system which holds the wound together and removes exudate and debris from the site to prevent infection. Dermabond is a surgical glue which holds the wound together to prevents infection. Prevena is more expensive to apply. However, the hypothesis is that the Prevena System will decrease infection rates and therefore, decrease the ultimate cost of the health care needed after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. In need of elective vascular procedure requiring ≥8 cm groin incision.
2. Able to provide consent
3. Able to care for wound or have support person to complete wound care
4. Willing to comply with follow-up

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2016-07; Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Harris, MD, Principal Investigator — State University of New York at Buffalo
Locations (2):
- United States (2):
  - Kaleida Health, Gates Vascular Institute, Buffalo, New York
  - State University of New York at Buffalo, Buffalo, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ploeg AJ, Lardenoye JW, Peeters MP, Hamming JF, Breslau PJ. Wound complications at the groin after peripheral arterial surgery sparing the lymphatic tissue: a double-blind randomized clinical trial. Am J Surg. 2009 Jun;197(6):747-51. doi: 10.1016/j.amjsurg.2008.04.014. Epub 2008 Oct 17. PMID 18929355
- [Background] Lee ES, Santilli SM, Olson MM, Kuskowski MA, Lee JT. Wound infection after infrainguinal bypass operations: multivariate analysis of putative risk factors. Surg Infect (Larchmt). 2000 Winter;1(4):257-63. doi: 10.1089/109629600750067183. PMID 12594881
- [Background] Lawlor DK, Derose G, Harris KA, Lovell MB, Novick TV, Forbes TL. The role of platelet-rich plasma in inguinal wound healing in vascular surgery patients. Vasc Endovascular Surg. 2011 Apr;45(3):241-5. doi: 10.1177/1538574411399157. PMID 21478245
- [Background] Exton RJ, Galland RB. Major groin complications following the use of synthetic grafts. Eur J Vasc Endovasc Surg. 2007 Aug;34(2):188-90. doi: 10.1016/j.ejvs.2007.03.012. Epub 2007 May 18. PMID 17512763
- [Background] Engin C, Posacioglu H, Ayik F, Apaydin AZ. Management of vascular infection in the groin. Tex Heart Inst J. 2005;32(4):529-34. PMID 16429897
- [Background] Bandyk DF. Vascular surgical site infection: risk factors and preventive measures. Semin Vasc Surg. 2008 Sep;21(3):119-23. doi: 10.1053/j.semvascsurg.2008.05.008. PMID 18774446
- [Background] Swinnen J, Chao A, Tiwari A, Crozier J, Vicaretti M, Fletcher J. Vertical or transverse incisions for access to the femoral artery: a randomized control study. Ann Vasc Surg. 2010 Apr;24(3):336-41. doi: 10.1016/j.avsg.2009.07.020. Epub 2009 Dec 4. PMID 19962270
- [Background] Dosluoglu HH, Loghmanee C, Lall P, Cherr GS, Harris LM, Dryjski ML. Management of early (<30 day) vascular groin infections using vacuum-assisted closure alone without muscle flap coverage in a consecutive patient series. J Vasc Surg. 2010 May;51(5):1160-6. doi: 10.1016/j.jvs.2009.11.053. Epub 2010 Mar 31. PMID 20356703
- [Background] Mangram AJ, Horan TC, Pearson ML, Silver LC, Jarvis WR. Guideline for prevention of surgical site infection, 1999. Hospital Infection Control Practices Advisory Committee. Infect Control Hosp Epidemiol. 1999 Apr;20(4):250-78; quiz 279-80. doi: 10.1086/501620. No abstract available. PMID 10219875
- [Background] Easterlin B, Bromberg W, Linscott J. A Novel Technique of Vacuum-assisted Wound Closure That Functions as a Delayed Primary Closure. Wounds. 2007 Dec;19(12):331-3. PMID 25942681
- [Background] de Lissovoy G, Fraeman K, Hutchins V, Murphy D, Song D, Vaughn BB. Surgical site infection: incidence and impact on hospital utilization and treatment costs. Am J Infect Control. 2009 Jun;37(5):387-397. doi: 10.1016/j.ajic.2008.12.010. Epub 2009 Apr 23. PMID 19398246
- [Background] Weir G. The use of a surgical incision management system on vascular surgery incisions: a pilot study. Int Wound J. 2014 Jun;11 Suppl 1(Suppl 1):10-2. doi: 10.1111/iwj.12261. PMID 24851730
- [Background] Matatov T, Reddy KN, Doucet LD, Zhao CX, Zhang WW. Experience with a new negative pressure incision management system in prevention of groin wound infection in vascular surgery patients. J Vasc Surg. 2013 Mar;57(3):791-5. doi: 10.1016/j.jvs.2012.09.037. Epub 2013 Jan 9. PMID 23312938
- [Background] Bruns TB, Worthington JM. Using tissue adhesive for wound repair: a practical guide to dermabond. Am Fam Physician. 2000 Mar 1;61(5):1383-8. PMID 10735344
- [Derived] Correia RM, Nakano LC, Vasconcelos V, Cristino MA, Flumignan RL. Prevention of infection in peripheral arterial reconstruction of the lower limb. Cochrane Database Syst Rev. 2025 Oct 29;10(10):CD015022. doi: 10.1002/14651858.CD015022.pub2. PMID 41159585
- [Derived] Cristino MA, Nakano LC, Vasconcelos V, Correia RM, Flumignan RL. Prevention of infection in aortic or aortoiliac peripheral arterial reconstruction. Cochrane Database Syst Rev. 2025 Apr 22;4(4):CD015192. doi: 10.1002/14651858.CD015192.pub2. PMID 40260835
- See also: Prevena TM Incision Management System — http://www.woundsource.com/product/prevena-incision-management-system

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from UBMD Vascular Surgery Office and were consented at the time of surgery at Buffalo General Medical Center between 2016 and 2019.
Period: Overall Study
Arm/Group | Prevena | Dermabond
Started | 50 | 55
Completed | 50 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Several patients randomized did not receive the randomized treatment based on physician decision, and were excluded from analysis as actual treatment rather than intent to treat was assessed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Prevena | Dermabond | Total
Number analyzed (Participants) | 46 | 55 | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 20 | 36
  >=65 years | 30 | 35 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (10) | 68 (12) | 68 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 15 | 36
  Male | 25 | 40 | 65
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 4 | 14
  White | 36 | 51 | 87
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 46 | 55 | 101

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Healing of Groin Wounds Between Patients Treated With Prevena vs Dermabond
Description: The primary effectiveness endpoint is 30 day healing of the randomized groin incision, with any wound infection or failure to heal. Szilagyi wound infection grade quantified on an ordinal scale will be used to assess the healing (None, Grade I: Infection contained to the dermis, Grade II: Infection extending into the subcutaneous tissue but the arterial graft is not involved, Grade III: Infection of the arterial graft or native vessel underlying the incision).
  Healing is assessed by complete sealing of the incision with no residual separation or drainage. All of the incisions were primarily closed, so a healed incision would have no gaps between the skin edges. This is a visual inspection.
  Szilagi is an assessment of the grade of wound infection for those that did not heal. It is well recognized and published, and noted as above for patients with vascular exposure.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Prevena | Dermabond
Number analyzed (Participants) | 46 | 55
Participants | 41 | 54

2. Secondary Outcome: Cost of Care
Description: Comparison of cost of treatment between the two arms
Time Frame: 30 days
Population: not analyzed as the primary outcome did not demonstrate improved outcomes, and the device being tested, wound vacuum, was more expensive. Had outcomes clinically been improved, financial assessment would have determined whether cost of infection outweighed cost of device.
Groups:
- Preveena: Outcome measures for cost were not calculated as initially planned as the primary outcome did not demonstrate any superiority with the Wound vacuum device, which is more expensive than the dermabond. Had there been improved clinical outcomes, financial benefit would have been assessed by comparing costs of infection vs device cost.
  As the primary outcome was not improved, this outcome was no longer necessary.
- Dermabond: Assessment not performed financially as Dermabond is less expensive than Preveena, and preveena did not achieve clinical superiority invalidating the need for this analysis to determine whether Preveena was more cost effective for the system.
Arm/Group | Preveena | Dermabond
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Visiting Nurses Home Visits and Physician Office Visits to Assess/Treat Wound Infection
Description: Physician office visits for diagnosis of Infection or visiting nurse visits for diagnosis of infection ONLY were assessed.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Prevena | Dermabond
Number analyzed (Participants) | 46 | 55
Participants | 7 | 7

ADVERSE EVENTS:
Time Frame: 40 days from time of surgery
Arm/Group | Prevena | Dermabond
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/55
Serious Adverse Events (participants affected / at risk) | 3/46 | 2/55
Other Adverse Events (participants affected / at risk) | 0/46 | 0/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prevena (N=46) | Dermabond (N=55)
Reoperation for groin complication (Infections and infestations) | 3 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2015-09-17): https://cdn.clinicaltrials.gov/large-docs/90/NCT02836990/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-08-11): https://cdn.clinicaltrials.gov/large-docs/90/NCT02836990/Prot_SAP_001.pdf